CLINICAL TRIAL: NCT01014702
Title: Prospective Clinical Trial of the LensAR Laser System in the Treatment of Cataracts of Different Grades of Maturity
Brief Title: Prospective Clinical Trial of the LensAR Laser System
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LensAR Incorporated (Industry)
Responsible Party: Keith Edwards, Director Clinical & Regulatory Affairs, LensAR Incorporated
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52-00006-000
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Cataract
Keywords: Cataract; Capsulotomy; Capsulorrhexis; lens fragmentation; phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Treatment (Experimental)
  Interventions: Device: LensAR Laser System
- Phacoemulsifcation (Active Comparator)
  Interventions: Device: Conventional phacoemulsification

INTERVENTIONS:
Device: LensAR Laser System — Use of laser for capsulotomy and lens fragmentation
  Arms: Laser Treatment
Device: Conventional phacoemulsification — Use of standard techniques for capsulotomy and lens fragmentation
  Arms: Phacoemulsifcation

SUMMARY:
The LensAR Laser System is used to create an opening in the anterior capsule of the lens and fragments the cataractous lens. The study will evaluate clinical outcomes compared to the contra-lateral eye treated with conventional phacoemulsification surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign and be given a copy of the written informed consent form
* Subjects must have elected to undergo lens extraction and IOL implantation and then elect to have the LensAR laser surgery as part of the procedure.
* Subjects must be willing and able to return for scheduled follow-up examinations for 6 months after surgery.
* Subjects must have central 7 mm of clear cornea without vascularization.

Exclusion Criteria:

* Subjects who have undergone previous corneal or intraocular surgery in the eye to be treated.
* Subjects with a history, signs or symptoms of ocular disease or atypical finding which would be contraindicated under standard of care for cataract surgery.
* Diabetic or hypertensive subjects with clinical evidence of retinal pathology.
* Subjects with macular degenerative pathology.
* Subjects with a history of steroid-responsive rise in IOP or uncontrolled glaucoma in either eye.
* Subjects with known lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Subjects with corneal disease or pathology that precludes applanation of the cornea or transmission of laser wavelength or distortion of laser light.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Completeness and ease of opening of capsulotomy | Day 0 (Surgery)
Reduced need for ultrasound phacoemulsification compared to control eye | Day 0 (surgery)
Rate of adverse events | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico IAP, Mexico City, Mexico